CLINICAL TRIAL: NCT04829968
Title: Valutazione Del Profilo di Emergenza e Del Sovracontorno in Corone Protesiche Complete su Denti Naturali Preparati Senza Linea di Finitura (BOPT): Studio Retrospettivo
Brief Title: Peri-implantitis in HIV-positive Patients
Acronym: PERIHIV2
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Luca Casula, MD, MSc resident in Oral Surgery, Università Vita-Salute San Raffaele
Other Study IDs: PERIHIV2
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; mucositis; HIV-positive patients; All-on-4
MeSH Terms: conditions — Peri-Implantitis; Mucositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: gingival conditions control — Peri-implant mucositis: It was diagnosed on the basis of the following criteria:
  1. Visual inspection demonstrating the following signs of inflammation in the peri-implant region: red as opposed to pink colour, swollen tissues as opposed to no swelling, and soft as opposed to firm tissue consistency.
  2. Presence of profuse (line or drop) bleeding and/or suppuration on probing.
  3. An increase in probing pocket depths (PPDs) compared to baseline. • Peri-implantitis: It was diagnosed on the basis of the following criteria:
  1. Visual inflammatory changes in the peri-implant soft tissues combined with bleeding on probing and/or suppuration.
  2. Increasing PPDs as compared to measurements recorded at the time of placement of supra-structures.

SUMMARY:
Objectives: This study aimed to assess the prevalence of peri-implantitis in human im-munodeficiency virus (HIV) -positive patients and the presence of a possible correlation between the immunological profile and serological values, of peri-implantitis, and of pos-sible differences between all-on-4 and single crown/bridge prostheses.

Subjects and methods: This retrospective study included 58 adult HIV-positive patients (222 implants) with either all-in-4 prostheses or single crowns/bridges on at least one dental implant loaded for more than a year who were followed for at least one year. Data pertaining to the probing pocket depth (PPD), bleeding on probing, and immunological and systemic profile were collected.

Results: Patients with single crown/bridge implant rehabilitation showed higher preva-lence of peri-implantitis (34%) than patients with all-on-4 rehabilitation (0%) (p=0.012). Patients with all-on-4 rehabilitation were significantly older than those with single crowns/bridges (p=0.004). Patients with peri-implantitis had implants for a significantly longer duration than those without (p=0.001), implying that the probability of peri-implantitis increases as the age of implant increases.

Conclusions: The prevalence of peri-implantitis was 26% in HIV-positive patients and 8% in dental implants. No correlation was found between patients' immunological and se-rological factors and peri-implantitis. The most important risk factor for peri-implantitis and mucositis was implant age.

DETAILED DESCRIPTION:
2.1 Type and sample of the study This retrospective monocentric observational study assessed the prevalence of peri-implant disease in HIV-positive patients treated at the department of dentistry of our hos-pital. At the same hospital, the HIV-positive patients were undergoing antiretroviral treat-ment. This study included 58 adult patients with at least one dental implant and a total of 222 implants followed for at least one year. Demographic, clinical, and laboratory infor-mation of the patients was collected. All procedures were approved by the appropriate lo-cal ethics committee. Appropriate informed consent forms were provided to all patients and were signed if the patients agreed to participate in the study.

This study has been reported according to the STrengthening the Reporting of OBserva-tional studies in Epidemiology (STROBE) guidelines and checklist.

2.2 Study design All included patients were divided into two groups, according to the type of prosthesis in-serted after implant placement (all-on-4 prosthesis versus single crowns\bridges), to as-sess the differences between the two types of prostheses in the inflammatory state, and therefore, in the presence of mucositis and peri-implantitis as well as in the variables ana-lysed.

As shown in Table 1, the data related to the immunological and systemic profile of the pa-tients (HIVRNA load, CD4+ level, CD8+ level, haemoglobin level, and platelet count) were collected through the database of the hospital.

2.3 Case definition for peri-implant condition: The clinical and radiological data for the diagnosis of peri-implant disease were collected according to the criteria laid in the Periodontology World Workshop in 2017 by Renvert et al. (2018).

2.3.1 Clinical Examination Data

* Peri-implant mucositis: It was diagnosed on the basis of the following criteria:

  1. Visual inspection demonstrating the following signs of inflammation in the peri-implant region: red as opposed to pink colour, swollen tissues as opposed to no swelling, and soft as opposed to firm tissue consistency.
  2. Presence of profuse (line or drop) bleeding and/or suppuration on probing.
  3. An increase in probing pocket depths (PPDs) compared to baseline.
* Peri-implantitis: It was diagnosed on the basis of the following criteria:

  1. Visual inflammatory changes in the peri-implant soft tissues combined with bleeding on probing and/or suppuration.
  2. Increasing PPDs as compared to measurements recorded at the time of placement of supra-structures.

     2.3.2 Radiological Examination Data Intraoral periapical radiographs are considered gold standard for radiological evaluation and were used in this study. The radiographic data were collected from the records of the patient. The position of the marginal bone was measured manually on an ultraspeed radio-graphic film (Ultra speed, Kodak, USA) using a dental calliper (0 to 10 mm). The distance to the marginal bone was measured from the mesial and distal aspects of the implants. The implant platform was used as a reference for the measurements. Two vertical lines were drawn parallel to a vertical line passing through the centre of the implant. The largest value was considered for statistical analysis. All assessments were performed by a single inves-tigator (LC).
* Peri-implantitis:

  1. Progressive bone loss in relation to the radiographic bone level assessment performed after one year following the delivery of the implant-supported prosthesis.

Inclusion criteria All patients (>18 years old), who were undergoing antiretroviral therapy at the same hos-pital, who had undergone prosthetic rehabilitation using one or more dental implants, with at least one year of follow-up after loading, and who had returned for a maintenance ap-pointment were considered for inclusion.

Exclusion criteria Patients who discontinued antiretroviral therapy, patients not undergoing therapy, patients whose previous radiographs and data on bleeding on probing and PPD at gingival level were unknown, patients with decompensated systemic diseases (for example, decompen-sated diabetes mellitus), patients treated with drugs that affect the bone turnover (for ex-ample, bisphosphonates), and patients under 18 years of age were not included in this study.

2.4 Statistical analysis A descriptive analysis was performed to assess all the obtained data. Continuous quantita-tive variables were described as medians and interquartile ranges, and categorical qualita-tive variables as frequencies and percentages (%). The continuous variables are graphical-ly represented using boxplots [the box shows the first (Q1), second (median), and third quartiles (Q3), and as whiskers, the values correspond to 1.5 times <Q1 and 1.5 times> Q3] and categorical variables using bar graphs. The quantitative variables were compared using the non-parametric Mann-Whitney test and qualitative variables using the chi-square test or Fisher's exact test. Stepwise multivariate logistic regression analysis was used to calculate the adjusted risks (odds), respective 95% confidence intervals, and probability (p-value) of developing peri-implantitis and mucositis. All analyses were performed using SAS for Windows Software (Version 9.4, SAS Institute). All statistical tests were ap-plied to 2 sails, and values were considered significant if the calculated probability was <0.05. The following two types of analyses were performed: the first analysed the varia-bles individually in the entire study population and the other in the population divided into 2 groups according to the type of implant-prosthetic rehabilitation performed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria All patients (>18 years old), who were undergoing antiretroviral therapy at the same hos-pital, who had undergone prosthetic rehabilitation using one or more dental implants, with at least one year of follow-up after loading, and who had returned for a maintenance ap-pointment were considered for inclusion.

Exclusion Criteria:

Exclusion criteria Patients who discontinued antiretroviral therapy, patients not undergoing therapy, patients whose previous radiographs and data on bleeding on probing and PPD at gingival level were unknown, patients with decompensated systemic diseases (for example, decompen-sated diabetes mellitus), patients treated with drugs that affect the bone turnover (for ex-ample, bisphosphonates), and patients under 18 years of age were not included in this study.

Age Groups: Child, Adult, Older Adult
Study Population: 58 HIV-positive patients
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Peri-implantitis prevalence | 3 years
  This study aimed to assess the prevalence of peri-implantitis in HIV-positive patients and to evaluate the presence of a possible correlation between the immunological profile and serological values of the same HIV-positive patients, of peri-implantitis, and of possible differences between all-on-4 and single crown/bridge prostheses in terms of peri-implant disease and the variables analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Casula, Monza, Monza E Della Brianza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casula L, Poli A, Clemente T, Artuso G, Cappare P, Gherlone EF. Prevalence of peri-implantitis in a sample of HIV-positive patients. Clin Exp Dent Res. 2021 Dec;7(6):1002-1013. doi: 10.1002/cre2.469. Epub 2021 Jul 20. PMID 34288560